CLINICAL TRIAL: NCT00356057
Title: AVAIL CLS/CRT: AV-node Ablation With CLS and CRT Pacing Therapies for the Treatment of AF
Brief Title: Investigational Device Exemption (IDE) Study for the Approval of Closed Loop Stimulation (CLS) and Cardiac Resyncronization Pacing Therapies (CRT) for the Treatment of Atrial Fibrillation (AF) With Ablate and Pace
Acronym: AVAIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G040150
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation; Congestive Heart Failure
Keywords: atrial fibrillation; AV node ablation; pacemaker; congestive heart failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Biventricular pacing group with Closed Loop Stimulation rate adaptation (Protos CLS device)
  Interventions: Device: Protos DR/CLS and Stratos LV CRT pacemakers
- 2 (Active Comparator): Biventricular pacing group with accelerometer based rate adaption (Stratos LV device)
  Interventions: Device: Protos DR/CLS and Stratos LV CRT pacemakers
- 3 (Active Comparator): Right Ventricular pacing group with accelerometer based rate adaption (Stratos LV device)
  Interventions: Device: Protos DR/CLS and Stratos LV CRT pacemakers

INTERVENTIONS:
Device: Protos DR/CLS and Stratos LV CRT pacemakers — Protos DR/CLS is a dual chamber pacemaker with CLS rate adaption, Stratos LV is a biventricular pacemaker with accelerometer based rate adaption
  Other Names: Protos DR/CLS dual chamber pacemaker

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of biventricular pacing over conventional right ventricular pacing in patients with persistent or permanent, symptomatic atrial fibrillation undergoing atrioventricular (AV) node ablation and permanent pacing therapy.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized, blinded trial. The study will consist of approximately 265 patients who require treatment of persistent or permanent, symptomatic atrial fibrillation by atrioventricular (AV) node ablation and permanent pacing therapy i.e. "Ablate and Pace" therapy. All patients enrolled into the clinical study will be randomly assigned to one of three groups using a randomization ratio of 2:2:1. Patients will be assigned to receive either biventricular (biV) pacing with CLS-based rate adaptive pacing using the legally marketed Protos DR/CLS (Group 1), or biventricular pacing with accelerometer-based rate adaptive pacing using the Stratos LV (Group 2), or right ventricular (RV) pacing with accelerometer-based rate adaptive pacing using the Stratos LV (Group 3). Patients in all three groups will be implanted with legally marketed right and left ventricular pacing leads. The patients, the core lab used to interpret the echocardiographic data and the Clinical Events Committee adjudicating crossover, patient death and congestive heart failure (CHF) hospitalizations will be blinded to the randomization assignment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for therapy
* Persistent, symptomatic AF with poorly controlled rapid ventricular rates or permanent, symptomatic AF with poorly controlled rapid ventricular rates.
* Eligible for AV nodal ablation and permanent pacemaker implantation
* NYHA Class II or III heart failure
* Age ≥ 18 years
* Understand the nature of the procedure
* Ability to tolerate the surgical procedure required for implantation
* Give informed consent
* Able to complete all testing required by the clinical protocol
* Available for follow-up visits on a regular basis at the investigational site

Exclusion Criteria:

* Meet one or more of the contraindications
* Have a life expectancy of less than six months
* Expected to receive heart transplantation within six months
* Enrolled in another cardiovascular or pharmacological clinical investigation
* Patients with an ICD, or being considered for an ICD
* Patients with previously implanted biventricular pacing systems
* Patients with previously implanted single or dual chamber pacing system with > 50% documented ventricular pacing
* Patients with previous AV node ablation
* Six-minute walk test distance greater than 450 meters
* Any condition preventing the patient from being able to perform required testing
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Conditions that prohibit placement of any of the lead systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Orlov, MD, Principal Investigator — Caritas Elizabeth, Boston, MA
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - Lake Charles Memorial, Lake Charles, Louisiana
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - St. Joseph Mercy, Ann Arbor, Michigan
  - McLaren Heart Foundation, Lapeer, Michigan
  - NYU Medical Center, New York, New York
  - Aultman Hospital, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Spartanburg Regional, Spartanburg, South Carolina
  - Lone Star Arrhythmia, Amarillo, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 153 patients were enrolled at 22 clinical sites from December 9, 2004 (the first implant of the study) through May 12, 2008.
Pre-assignment Details: No patients were excluded before assigment to groups. A total of 27 patients did not receive a device implant due to withdrawal of consent, inelegibility after randomization and unability to implant the LV lead.
Groups:
- biV-pacing With CLS Rate Adaption (Protos CLS): Patients are implanted with a Protos CLS device, using the atrial port of the device for the left ventricular lead and the ventricular port for the ventricular lead to provide biV pacing. CLS is activated for rate adaptation.
- biV Pacing With Accelerometer Based Rate Adaption (Stratos LV): Patients are implanted with a Stratos LV device, with the atrial port plugged and the left ventricular port for the left ventricular lead and the right ventricular port for the right ventricular lead to provide biV pacing. The acceleromer is activated for rate adaptation.
- RV Pacing With Accelerometer Based Rate Adaption (Stratos LV): Patients are implanted with a Stratos LV device, with the atrial port plugged and the left ventricular port for the left ventricular lead and the right ventricular port for the right ventricular lead to provide biV pacing. The device is programmed to right ventricular pacing only. The acceleromer is activated for rate adaptation.
Period: Overall Study
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Started | 58 | 61 | 34
IMPLANTED | 49 | 52 | 25
Completed | 45 | 47 | 22
Not Completed | 13 | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | Total
Number analyzed (Participants) | 58 | 61 | 34 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.4) | 72.7 (7.8) | 72.3 (8.2) | 73.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 17 | 90
  Male | 24 | 22 | 17 | 63
Region of Enrollment [Number; unit: participants]
  United States | 57 | 59 | 33 | 149
  Canada | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Percentage Improvement From Baseline of the 6-minute Walk Test Distance and Minnesota Living With Heart Failure Quality of Life Score at 6-months
Description: Combined, average percentage improvement in 6-minute walk test distance and Minnessota Living With Heart Failure Quality of Life score from baseline to 6-month follow-up for the Protos DR/CLS (Group 1) and Stratos LV (Group 2) compared with the active control (Group 3). The 6-minute walk test is a test that measure how far a patient can walk in 6 minutes in a standardized walking course. Percent Change (0% (worst)-100% (best))
Time Frame: Change from baseline to six months post-procedure
Population: Patients included in this analysis are those patients with complete six minute walk test and Quality of Life data at both baseline and the six-month follow-up.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 43 | 43 | 22
Percent Change | 40.1 (5.7) | 42.5 (8.9) | 31.5 (9.0)
Statistical Analysis 1: Comparison: biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.437, t-test, 2 sided
Statistical Analysis 2: Comparison: biV-pacing With CLS Rate Adaption (Protos CLS) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.405, t-test, 2 sided

2. Primary Outcome: Number of Participants Free of System-related Complications (Related to the Device, Leads, or Implant Procedure) at 6 Months Post-procedure
Description: Complication-free rate was evaluated in an equivalence (non-inferiority) format compared to a target of 85% minus delta (10%), where delta is the clinically significant difference for establishing equivalence. This endpoint evaluated system-related complications.
Time Frame: At six months post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Protos DR/CLS System: Protos DR/CLS (biV pacing with CLS rate adaptation)
Arm/Group | Protos DR/CLS System
Number analyzed (Participants) | 58
Participants | 49
Statistical Analysis 1: Comparison: Protos DR/CLS System; Test type: Equivalence — Complication-free rate was evaluated in an equivalence (non-inferiority) format compared to a target of 85% minus delta (10%), where delta is the clinically significant difference for establishing equivalence; p = 0.0596, t-test, 1 sided

3. Primary Outcome: Number of Participants Free of System-related Complications (Related to the Device, Leads, or Implant Procedure) at 6 Months Post-procedure
Description: Complication-free rate was evaluated in an equivalence (non-inferiority) format compared to a target of 85% minus delta (10%), where delta is the clinically significant difference for establishing equivalence. This endpoint evaluated system-related complications. All Stratos systems (in both the biV and RV pacing arms) were evaluated together as pre-specified in the protocol.
Time Frame: At six months post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Stratos LV System: Stratos LV (biV or RV pacing groups with accelerometer based rate adaptation)
Arm/Group | Stratos LV System
Number analyzed (Participants) | 95
Participants | 84
Statistical Analysis 1: Comparison: Stratos LV System; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0009, t-test, 1 sided

4. Secondary Outcome: Change in Six-minute Walk Test
Time Frame: Change from baseline to 6 months post-procedure
Population: Subjects with paired baseline and 6-month six-minute walk test data.
Measure: Mean (Standard Error); unit: Meters
Groups:
- biV-pacing With CLS Rate Adaption (Protos CLS): Biventricular pacing group with Closed Loop Stimulation rate adaptation (Protos CLS device)
- biV Pacing With Accelerometer Based Rate Adaption (Stratos LV): Biventricular pacing group with accelerometer based rate adaption (Stratos LV device)
- RV Pacing With Accelerometer Based Rate Adaption (Stratos LV): Right Ventricular pacing group with accelerometer based rate adaption (Stratos LV device)
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 44 | 44 | 22
Meters | 48.1 (13.2) | 49.3 (12.9) | 54.5 (20.9)

5. Secondary Outcome: Change in Quality Of Life (QOL) Score Over 6 Months Calculated as QOL Score at Baseline - QOL Score at 6 Months
Description: Quality of Life was evaluated using the Minnesota Living with Heart Failure (MLHF) Quality of Life (QOL) Questionnaire.The questionnaire consists of 21 questions to measure the subjects' perception of how their HF and its treatment affected their ability to live as they wanted during the last month. The questions describe different ways in which some people are affected (i.e. physical, socioeconomic, and psychological impairments). If a question does not apply to a subject or is not related to their HF, then they can answer with a 0. If it does apply to them, then they can rate (from 1 to 5) how much it has affected them. From the 21 questions, the lowest possible total score is 0, and the highest possible total score is 105. A lower score is desirable. This outcome was calculated as QOL score at baseline minus QOL score at 6 months. Therefore, a positive change in QOL score represents an improvement in quality of life, while a negative change in QOL score represents a worsening.
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month QOL data. A positive score represents improvement from baseline to 6-months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 43 | 45 | 22
units on a scale | 28.9 (3.9) | 25.2 (3.2) | 24.5 (6.1)

6. Secondary Outcome: Cardiac Remodeling Assessments by Echocardiography - Change in Left Ventricular Ejection Fraction
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month echocardiography data.
Measure: Mean (Standard Error); unit: percent
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 36 | 42 | 14
percent | 3.1 (1.3) | 3.4 (0.9) | -2.6 (2.6)
Statistical Analysis 1: Comparison: biV-pacing With CLS Rate Adaption (Protos CLS) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.030, t-test, 2 sided
Statistical Analysis 2: Comparison: biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.006, t-test, 2 sided

7. Secondary Outcome: Changes in New York Heart Association (NYHA) Classification
Description: The purpose is to evaluate the change in the participant's NYHA classification.
  There are four NYHA classes:
  Class I: Patients with cardiac disease, but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month NYHA classification data. The outcome of "Improved at least 1 Class" represents a numerically higher NYHA class at baseline than at 6 months (e.g. NYHA class III at baseline changed to NYHA class II at 6 months).
Measure: Count of Participants; unit: Participants
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 44 | 45 | 22
Participants
  Improved at least 1 Class | 24 | 26 | 9
  No change | 17 | 17 | 11
  Worsened at least 1 Class | 3 | 2 | 2

8. Secondary Outcome: Percentage of Patients With Congestive Heart Failure (CHF) Related Hospitalizations
Time Frame: At six months post-procedure
Population: Subjects successfully implanted with investigational system.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 49 | 52 | 25
percentage of participants analyzed | 20 | 13 | 16

9. Secondary Outcome: Mortality Rate
Time Frame: At six months post-procedure
Population: Subjects enrolled
Measure: Number; unit: percentage of participants analyzed
Groups:
- biV-pacing With CLS Rate Adaption (Protos CLS): Biventricular pacing group with CLS rate adaptation (Protos CLS device)
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 58 | 61 | 34
percentage of participants analyzed | 1.7 | 11.5 | 5.9

10. Secondary Outcome: Cardiac Remodeling Assessments by Echocardiography - Change in Left Atrial Volume
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month echocardiography data.
Measure: Mean (Standard Error); unit: mL
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 37 | 41 | 18
mL | -3.2 (2.8) | -1.1 (2.8) | 13.7 (6.0)
Statistical Analysis 1: Comparison: biV-pacing With CLS Rate Adaption (Protos CLS) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.014, t-test, 2 sided

11. Secondary Outcome: Cardiac Remodeling Assessments by Echocardiography - Change in Left Ventricular Mass
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month echocardiography data.
Measure: Mean (Standard Error); unit: grams
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 41 | 45 | 19
grams | -1.2 (5.7) | -14.5 (8.3) | 25.1 (10.5)
Statistical Analysis 1: Comparison: biV-pacing With CLS Rate Adaption (Protos CLS) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.020, t-test, 2 sided
Statistical Analysis 2: Comparison: biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.008, t-test, 2 sided

12. Secondary Outcome: Cardiac Remodeling Assessments by Echocardiography - Change in Left Ventricular End Systolic Volume
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month echocardiography data.
Measure: Mean (Standard Error); unit: mL
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 36 | 42 | 15
mL | -7.7 (1.7) | -5.9 (2.1) | 8.7 (4.6)
Statistical Analysis 1: Comparison: biV-pacing With CLS Rate Adaption (Protos CLS) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.001, t-test, 2 sided

13. Secondary Outcome: Cardiac Remodeling Assessments by Echocardiography - Change in Left Ventricular End Diastolic Volume
Time Frame: Change from baseline to six months post-procedure
Population: Subjects with paired baseline and 6-month echocardiography data.
Measure: Mean (Standard Error); unit: mL
Arm/Group | biV-pacing With CLS Rate Adaption (Protos CLS) | biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) | RV Pacing With Accelerometer Based Rate Adaption (Stratos LV)
Number analyzed (Participants) | 36 | 42 | 15
mL | -10.1 (3.5) | -7.1 (4.0) | 9.5 (8.2)
Statistical Analysis 1: Comparison: biV-pacing With CLS Rate Adaption (Protos CLS) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.039, t-test, 2 sided
Statistical Analysis 2: Comparison: biV Pacing With Accelerometer Based Rate Adaption (Stratos LV) vs RV Pacing With Accelerometer Based Rate Adaption (Stratos LV); Test type: Superiority; p = 0.047, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Study duration with a mean enrollment duration of 19.6 months.
Description: Adverse events are included for all study groups together.
Arm/Group | All Groups
All-Cause Mortality (participants affected / at risk) | 10/153
Serious Adverse Events (participants affected / at risk) | 58/153
Other Adverse Events (participants affected / at risk) | 102/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Groups (N=153)
Device related (Cardiac disorders) | 4 (5)
LV lead related (Cardiac disorders) | 10 (10)
Other medical (Cardiac disorders) | 45 (65)
Procedure (Cardiac disorders) | 4 (4)
RV-lead related (Cardiac disorders) | 9 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Groups (N=153)
LV lead related (Cardiac disorders) | 30 (30)
RV lead related (Cardiac disorders) | 2 (2)
Device related (Cardiac disorders) | 12 (12)
Procedure (Cardiac disorders) | 48 (53)
Other medical (Cardiac disorders) | 55 (90)

LIMITATIONS AND CAVEATS:
Early termination due lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.